CLINICAL TRIAL: NCT04223804
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1b Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of ABBV-181 in HIV-1 Infected Adults
Brief Title: A Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of ABBV-181 (Budigalimab) in Adult Participants With Human Immunodeficiency Virus (HIV)-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M19-939; 2019-004866-16 (EudraCT Number)
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Human Immunodeficiency Virus (HIV); HIV Infection; HIV-1
Keywords: Human Immunodeficiency Virus (HIV); HIV Infection; HIV-1; ABBV-181; Analytical Treatment Interruption; Budigalimab; Programmed cell death protein-1 (PD-1); Anti-PD-1 Antibody
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — budigalimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Stage 1: Arm A (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo
- Stage 1: Arm B (Experimental): Participants will receive ABBV-181 dose A.
  Interventions: Drug: ABBV-181
- Stage 1: Arm C (Experimental): Participants will receive ABBV-181 dose B.
  Interventions: Drug: ABBV-181
- Stage 2: Arm D (Placebo Comparator): Participants will receive Placebo.
  Interventions: Drug: Placebo
- Stage 2: Arm E (Experimental): Participants will receive ABBV-181 dose C.
  Interventions: Drug: ABBV-181

INTERVENTIONS:
Drug: ABBV-181 — Intravenous (IV) Infusion
  Other Names: Budigalimab
  Arms: Stage 1: Arm B; Stage 1: Arm C; Stage 2: Arm E
Drug: Placebo — Intravenous (IV) infusion
  Arms: Stage 1: Arm A; Stage 2: Arm D

SUMMARY:
This study will be conducted in two stages and will test the safety/tolerability, pharmacokinetics (how the body handles study drug) and pharmacodynamics (effects on the immune system and the virus) of the study drug ABBV-181 in Human immunodeficiency virus (HIV)-1 infected participants undergoing Antiretroviral therapy (ART) interruption.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 18.0 and 35 kg/m2.
* HIV-1 infected on antiretroviral therapy (ART) for at least 12 months prior to screening and on current ART regimen for at least 8 weeks prior to screening.
* Meets HIV-specific laboratory parameters as below:

  * Plasma HIV-1 RNA below lower limit of quantification (LLOQ) at screening and at least 6 months prior to screening.
  * CD4+ T cell count >= 500 cells/uL at screening and at least once during the 12 months prior to screening.
  * CD4+ T cell nadir of >= 200 cells/uL during chronic infection.
* Willing to undergo ART interruption.
* Agrees to use an effective barrier method of protection (male and/or female condoms) during sexual activity for protection against HIV-1 transmission throughout the entire study.

Exclusion Criteria:

* Known resistance to at least 2 classes of ART.
* History of AIDS-defining illness.
* Active or suspected malignancy or history of malignancy (other than basal cell skin cancer or cervical carcinoma in situ) in the past 5 years.
* History of or active immunodeficiency (other than HIV).
* Active autoimmune disease or history of autoimmune disease that has required systemic treatment.
* Prior receipt of immunomodulatory or immunosuppressive (including intravenous infusion or oral steroids at any dose, but excluding steroids that are inhaled, topical or by local injection) therapy within 24 weeks prior to the first dose of study drug.
* Prior therapy/exposure to ABBV-181 or any other immune checkpoint inhibitor.
* Current hepatitis B virus or hepatitis C virus infection.
* Clinically significant medical disorders that might expose the participants to undue risk of harm, confound study outcomes, or prevent the participant from completing the study (including but not limited to significant or unstable cardiac, neurologic or pulmonary disease, chronic active infectious disease except for HIV, chronic liver disease, poorly controlled diabetes mellitus and history of Stevens Johnson Syndrome toxic epidermal necrolysis (TEN), or drug reaction with eosinophilia and systemic symptoms (DRESS)).
* Known psychiatric or substance abuse disorders that would interfere with adherence to study requirements.
* Female participants must not be pregnant, breastfeeding, or considering becoming pregnant during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Study Drug-Related Adverse Events Grade 3 or Higher | Up to approximately 44 weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of the study drug as either having a reasonable possibility or no reasonable possibility. AEs are given a grade from 1-5 with Grade 3 being severe but not life-threatening and requiring hospitalization, Grade 4 being life-threatening requiring immediate intervention and Grade 5 being death related to an AE.
Number of Participants with Study Drug-Related Immune-Related Adverse Events (IRAE) | Up to approximately 44 weeks
  Assessed using the American Society of Clinical Oncology (ASCO) IRAE management guidelines (which utilizes the NIH CTCAE grading scale) but modified, as applicable, according to the NIH Division of AIDS (DAIDS) (v2.1) AE grading scale.
Number of Participants with Adverse Events (AEs) Corresponding to Retroviral Rebound Syndrome | Up to approximately 44 weeks
  Adverse Events (AEs) Corresponding to Retroviral Rebound Syndrome.
Maximum Observed Concentration (Cmax) | Up to approximately 36 weeks
  Maximum Observed Concentration (Cmax) of ABBV-181.
Time to Cmax (Tmax) | Up to approximately 36 weeks
  Time to Cmax (Tmax) of ABBV-181.
Observed Concentration (Ctrough) | Up to approximately 36 weeks
  Observed Concentration (Ctrough) at the end of the dosing intervals for ABBV-181.
Area Under the Curve (AUCtau) | Up to approximately 36 weeks
  Area Under the Curve (AUCtau) during the dosing intervals for ABBV-181.
Half-life (t1/2) | Up to approximately 36 weeks
  Half-life (t1/2) of ABBV-181 following the last dose.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (23):
- United States (15):
  - Franco Felizarta, Md /Id# 215721, Bakersfield, California
  - Ruane Clinical Research Group /ID# 224866, Los Angeles, California
  - Quest Clinical Research /ID# 215796, San Francisco, California
  - George Washington University Medical Faculty Associates /ID# 213893, Washington D.C., District of Columbia
  - Midway Immunology and Research /ID# 215587, Ft. Pierce, Florida
  - University of Miami, Miller School of Medicine /ID# 213833, Miami, Florida
  - Orlando Immunology Center /ID# 243276, Orlando, Florida
  - Triple O Research Institute /ID# 224863, West Palm Beach, Florida
  - Be Well Medical Center /ID# 223841, Berkley, Michigan
  - Mayo Clinic - Rochester /ID# 217820, Rochester, Minnesota
  - Saint Michael's Medical Center /ID# 228733, Newark, New Jersey
  - University of Cincinnati /ID# 215615, Cincinnati, Ohio
  - Prism Health North Texas - Oak Cliff Health Center /ID# 214036, Dallas, Texas
  - North TX Infectious Diseases /ID# 224861, Dallas, Texas
  - Peter Shalit, M.D. /ID# 224870, Seattle, Washington
- Australia (3):
  - Holdsworth House Medical Practice /ID# 215352, Darlinghurst, New South Wales
  - St Vincent's Hospital Sydney /ID# 215354, Darlinghurst, New South Wales
  - The Royal Melbourne Hospital /ID# 215351, Parkville, Victoria
- Canada (3):
  - Ottawa Hospital Research Institute /ID# 218083, Ottawa, Ontario
  - Toronto General Hospital /ID# 218082, Toronto, Ontario
  - McGill Univ Clinical Research /ID# 218081, Montreal, Quebec
- Puerto Rico (2):
  - Clinical Research Puerto Rico /ID# 218821, San Juan
  - Puerto Rico AIDS Clinical Trials Unit CRS /ID# 213761, San Juan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramgopal MN, Lalezari JP, Pires Dos Santos AG, Krishnan P, Vaidya TR, Zhou F, Betman H, Dorr P, Mostafa NM, Alcaide ML, Felizarta F, Routy JP. Budigalimab, an anti-PD-1 inhibitor, for people living with HIV-1: a randomized, placebo-controlled phase 1b study. Nat Med. 2025 Nov;31(11):3879-3888. doi: 10.1038/s41591-025-03993-0. Epub 2025 Oct 15. PMID 41094034